CLINICAL TRIAL: NCT02408887
Title: Randomized Controlled Trial of Total Thyroidectomy With and Without Prophylactic Central Neck Lymph Node Dissection in Patients With Low-risk Papillary Thyroid Cancer
Brief Title: Total Thyroidectomy With and Without Prophylactic Central Neck Lymph Node Dissection in People With Low-risk Papillary Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Naris Nilubol, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150105; 15-C-0105
Record Dates: First submitted 2015-04-03; First posted 2015-04-06 (Estimated); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Low-risk Papillary Thyroid Cancer; Endocrine Malignancy; Thyroid Cancer
Keywords: Thyroidectomy; Serum Thyroglobulin; Quality of Life; Central Neck Lymph Node Metastasis; Central Neck Lymph Node Dissection
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) (Active Comparator): TT plus pCND
  Interventions: Procedure: Total Thyroidectomy (TT); Procedure: Prophylactic central neck lymph node dissection (pCND)
- Arm 1/Total Thyroidectomy (TT) alone (Active Comparator): TT alone
  Interventions: Procedure: Total Thyroidectomy (TT)

INTERVENTIONS:
Procedure: Total Thyroidectomy (TT) — Total removal of thyroid
Procedure: Prophylactic central neck lymph node dissection (pCND) — Lymph node dissection
  Arms: Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND)

SUMMARY:
Background:

- Papillary thyroid cancer (PTC) often spreads to lymph nodes in the neck. This can be hard to detect. People often have lymph nodes removed anyway, and researchers want to study if this is a good idea.

Objective:

- To compare the effectiveness of removing lymph nodes in the neck that show no evidence of cancer along with the thyroid, or removing only the thyroid.

Eligibility:

- Adults age 18 and older with PTC or thyroid nodules suspicious for PTC, with no evidence that the disease has spread in the body.

Design:

* Participants will be screened with medical history, physical exam, blood tests, scans, and x-rays.
* Participants will:
* Answer questions. They may have a tumor biopsy.
* Have a flexible laryngoscopy. A small tube will pass through the nose to the vocal cords.
* Group 1: have surgery to remove the thyroid gland only. Lymph nodes in the neck will be removed if the cancer has spread.
* Group 2: have surgery to remove the thyroid and lymph nodes in the neck.
* At all post-surgery visits, participants will answer questions and have blood drawn. In addition:
* 1 day: laryngoscopy.
* 2 weeks: possible laryngoscopy.
* 3 months: ultrasound of the thyroid and neck.
* Discuss whether to try hormone treatment and/or radioactive iodine.
* Possible diagnostic whole body radioiodine scan (WBS). Participants will swallow a capsule or liquid and lie under a camera.
* 6 months: ultrasound and maybe laryngoscopy.
* 1 year: diagnostic WBS and ultrasound. Participants may get thyroid stimulating hormone.
* Participants will have annual follow-up visits for 10 years. They will have a physical exam, blood drawn, scans, and may complete a questionnaire.

DETAILED DESCRIPTION:
Background:

* Thyroid cancer is the most common endocrine malignancy and papillary thyroid cancer (PTC) accounts for more than 80% of thyroid cancer.
* The incidence of thyroid cancer has risen over the past decades.
* Central neck lymph node metastasis (LNM) is common in PTC and preoperative imaging studies do not identify all involved lymph nodes in the central neck.
* It remains controversial if prophylactic central neck lymph node dissection (pCND) in patients with low-risk PTC results in lower rates of persistent/recurrent disease and higher complication rates as there has been no randomized controlled trial addressing these issues to date.
* Serum thyroglobulin (Tg), especially when thyroid stimulating hormone (TSH)-stimulated, is a very sensitive and specific marker for persistent/recurrent PTC, in the absence of interfering anti-Tg antibodies.
* Retrospective studies have compared the postoperative TSH-stimulated Tg levels between those who underwent prophylactic central neck dissection (pCND) and those who did not with conflicting results. A randomized trial is needed.
* Health-related quality of life (QOL) is a well-accepted tool to measure the outcome of cancer treatments. Short-form 36 (SF-36) version 2 (v2) questionnaire has been frequently used to evaluate the QOL in patients with thyroid cancer. There is no study evaluating the difference in QOL in patients with low-risk PTC undergoing total thyroidectomy (TT) with and without pCND.

Objectives:

-To determine and compare biochemical cure rates in patients with low-risk PTCs undergoing total thyroidectomy (TT) with and without pCND as measured by postoperative TSH-stimulated serum thyroglobulin (stim-Tg) at 3 months (prior to radioactive iodine treatment (RAI) treatment).

Eligibility:

* Patients greater than or equal to 18 years who have thyroid nodule(s) greater than or equal to 1 cm. but less than or equal to 4 cm. in size with either:

  * inconclusive thyroid cytology positive for B-Raf Proto-oncogene Serine/Threonine Kinase (BRAF) Valine 600 Glutamic Acid (V600E) mutation or rearranged in transformation/papillary thyroid carcinomas (RET/PTC) rearrangement or
  * cytologically suspicious for or consistent with PTC
* Absence of extrathyroidal extension or lymphadenopathy suggesting metastatic PTC on physical examination and neck ultrasound.

Design:

* Prospective, single-blinded, randomized controlled clinical trial.
* Cytology will be reviewed by Laboratory of Pathology, National Cancer Institute (NCI) or a pathology laboratory at the enrolling institution. Once patients provide written informed consent, they will receive routine history, physical, radiographic (neck ultrasonography (USG), and/or other indicated tests) examinations as well as blood tests. Preoperative fine needle aspiration for cytology and BRAFV600E mutation will be performed if participant has not had either test performed.
* Preoperative assessment of QOL using standardized questionnaire (SF-36 v2) will be obtained within 30 days prior to surgery
* Preoperative vocal cord assessment will be done by flexible laryngoscopy.
* Participants will be randomized after clinical staging, including ultrasonography, to receive TT and pCND or TT alone and will be blinded from the result of randomization and treatment. Patients will remain blinded from treatment assignment for the duration of the study except for patients assigned to TT alone but found to have lymph node metastases as described below.
* If participants in TT alone group are found to have lymph node metastasis at the time of the operation by frozen section analysis, a therapeutic central neck dissection (CND) will be performed. Participants will remain in the intention to treat (TT alone) group. TT patients will be informed if a therapeutic CND is indicated and as such the blind will be broken for these patients prior to study completion.
* All participants will have intact parathyroid hormone (PTH), calcium and electrolytes checked preoperatively, in the morning after surgery, 2 weeks, and 6 months postoperatively.
* Postoperative flexible laryngoscopy will be performed on postoperative day 1 (or postoperative day 2, if it cannot be performed on the first postoperative day) and 6 months postoperatively if vocal cord abnormality is found on postoperative day 1
* Postoperative assessment of QOL will be done on day 1, 2 weeks, 3 months and 6 months, 1, 5 and 10 years postoperatively.
* Participants with postoperative hypoparathyroidism (low PTH and hypocalcemia) will be treated with calcium replacement with or without vitamin D analogue. Serum PTH and electrolytes will be monitored until resolved.
* Stim-Tg will be checked at 3 months postoperatively (prior to RAI scan/ablation, if indicated) and at 1 year postoperatively or 1 year post-remnant ablation. 1 year stim-Tg evaluation will be performed in patients enrolled at the NIH but is optional in patients enrolled at non-NIH site(s) Unstimulated Tg, thyroid function tests, and anti-thyroglobulin antibodies will be checked annually for 10 years.
* Soft tissue neck ultrasonography will be performed in all patients preoperatively and every year postoperatively for the first 10 years.
* If biochemical evidence of tumor recurrence occurs, patients will undergo appropriate radiographic studies and/or nuclear scintigraphy. Tissue biopsy of suspicious lesion(s) will be performed if clinically indicated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed at least 1 thyroid nodule that is greater than or equal to1 cm. but less than or equal to 4 cm measured in greatest dimension and confirmed by the Laboratory of Pathology, National Cancer Institute (NCI) or confirmed by the pathology laboratory of the enrolling institution:

  * Indeterminate thyroid biopsy per Bethesda System for reporting thyroid cytopathology with B-Raf Proto-oncogene Serine/Threonine Kinase (BRAF) Valine 600 Glutamic Acid (V600E) mutation or rearranged in transformation/papillary thyroid carcinomas (RET/PTC) rearrangement
  * Cytologically or histologically suspicious or confirmed PTC per Bethesda System for reporting thyroid cytopathology.
* Age greater than or equal to 18 years. Because PTC occurs rarely in patients <18 years of age, children are excluded from this study.
* Absence of radiographic evidence of extrathyroidal extension.
* Absence of abnormal lymphadenopathy suggesting metastatic PTC on physical examination and/or imaging studies.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients must have adequate organ function to safely undergo general anesthesia and thyroidectomy. Laboratory values obtained less than or equal to 4 weeks prior to surgery must demonstrate adequate bone marrow function (hemoglobin (Hb) greater than or equal to 6.0 mmol/L, absolute neutrophil count greater than or equal to 1.5 x 10^9/L, platelets greater than or equal to 80 x 10^9/L), liver function (serum bilirubin less than or equal to 2 x upper limit of normal (ULN), serum transaminases less than or equal to 3 x ULN). Patients with chronic kidney disease who are on chronic renal replacement therapy are allowed. Other tests, such as pulmonary function tests, cardiac echocardiogram or stress test, will be performed if clinically indicated.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Women must not become pregnant prior to surgery or during the first 3 months after surgery. Women who can become pregnant will be asked to practice an effective form of birth control for up to 3 months after surgery.

EXCLUSION CRITERIA:

* Patients who have had previous thyroid surgery
* Patients whose tumors are deemed unresectable by clinical/imaging criteria.
* Patients with known synchronous distant metastatic disease.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded because we do not want to expose the unborn child to the procedures necessary to perform the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded, linked data in a National Institutes of Health (NIH)-funded or approved public repository. Coded, linked data in Biomedical Translational Research Information System (BTRIS) (automatic for activities in the Clinical Center). Identified or coded, linked data with approved participating sites under appropriate agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before publication. At the time of publication or shortly thereafter.
Access Criteria: A National Institutes of Health (NIH)-funded or approved public repository, clinicaltrials.gov. Biomedical Translational Research Information System (BTRIS) (automatic for activities in the Clinical Center). Publication and/or public presentations.

REFERENCES:
- [Background] Lang BH, Wong KP, Wan KY, Lo CY. Significance of metastatic lymph node ratio on stimulated thyroglobulin levels in papillary thyroid carcinoma after prophylactic unilateral central neck dissection. Ann Surg Oncol. 2012 Apr;19(4):1257-63. doi: 10.1245/s10434-011-2105-5. Epub 2011 Oct 12. PMID 21989667
- [Background] Iyer NG, Morris LG, Tuttle RM, Shaha AR, Ganly I. Rising incidence of second cancers in patients with low-risk (T1N0) thyroid cancer who receive radioactive iodine therapy. Cancer. 2011 Oct 1;117(19):4439-46. doi: 10.1002/cncr.26070. Epub 2011 Mar 22. PMID 21432843
- [Background] Lee J, Kwon IS, Bae EH, Chung WY. Comparative analysis of oncological outcomes and quality of life after robotic versus conventional open thyroidectomy with modified radical neck dissection in patients with papillary thyroid carcinoma and lateral neck node metastases. J Clin Endocrinol Metab. 2013 Jul;98(7):2701-8. doi: 10.1210/jc.2013-1583. Epub 2013 May 15. PMID 23678034
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0105.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND): pCND plus TT
  Total Thyroidectomy (TT): Total removal of thyroid
  Prophylactic central neck lymph node dissection (pCND): Lymph node dissection
Period: Overall Study
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Started | 8 | 6
Completed | 7 | 5
Not Completed | 1 | 1
Not completed — Participant was inevaluable due to advanced cancer | 1 | 0
Not completed — Participant was inevaluable due to benign pathology. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (14.35) | 56.17 (14.16) | 48.93 (15.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1
  White | 5 | 4 | 9
  Asian | 0 | 1 | 1
  Hispanic | 3 | 2 | 5
  Non-Hispanic | 5 | 4 | 9
  Unknown | 1 | 1 | 2
  Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Have Biochemical Cure After Total Thyroidectomy (TT) With and Without Prophylactic Central Neck Lymph Node Dissection (pCND)
Description: number of participants that have biochemical cure after total thyroidectomy (TT) with and without pCND as measured by postoperative thyroid stimulating hormone (TSH)-stimulated serum thyroglobulin (stim-Tg). Per protocol, Biochemical cure is defined as "stim-Tg < 2 ng/ml or unstimulated Tg ≤ 0.2 ng/ml" post-surgery. Biochemical persistent or recurrent disease is suspected when stim-Tg ≥5 ng/ml or unstimulated Tg >0.3 ng/ml or a conversion or a rise in anti-Tg antibodies.
Time Frame: At 3 months (prior to radioactive iodine (RAI) treatment)
Population: One participant in Arm 2, and two participants in Arm 1 was inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 4
Participants
  Biochemical cure | 7 | 3
  Biochemical persistent or recurrent disease | 0 | 1

2. Secondary Outcome: Number of Participants That Have Biochemical Cure After Total Thyroidectomy (TT) With and Without Prophylactic Central Neck Lymph Node Dissection (pCND)
Description: Participants that have biochemical cure after TT with and without pCND by postoperative thyroid-stimulating hormone (TSH)-stimulated serum thyroglobulin (stim-Tg) at 1 year postoperatively in participants who will not receive radioactive iodine (RAI) or 1 year post remnant ablation. Per protocol, Biochemical cure is defined as "stim-Tg < 2 ng/ml or unstimulated Tg ≤ 0.2 ng/ml" post-surgery. Biochemical persistent or recurrent disease is suspected when stim-Tg ≥5 ng/ml or unstimulated Tg >0.3 ng/ml or a conversion or a rise in anti-Tg antibodies.
Time Frame: Up to 1 year postoperatively or 1 year post remnant ablation.
Population: One participant in Arm 2, and two participants in Arm 1 was inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 4
Participants
  Biochemical cure | 6 | 4
  Biochemical persistent or recurrent disease | 0 | 0
  Inconclusive evidence of biochemical cure | 1 | 0

3. Secondary Outcome: Number of Participants Who Completed Quality of Life (QOL) Survey at Following Timepoints: Quality of Life After Total Thyroidectomy (TT) With and Without Prophylactic Central Neck Lymph Node Dissection (pCND)
Description: Number of participants that completed the Quality-of-Life SF-36 questionnaire after TT with and without pCND.
Time Frame: pre-operation(op), post-op day 1 and 2, 2 and 3 weeks post-op, 3, 6 and 9 months post-op, 1 and 2 years post-op. Approximately 4 years.
Population: Not all participants in the respective Arms had completed SF-36 surveys in the timepoints stated in the protocol. The SF-36 survey responses were not scored prior to closure of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
Participants
  Pre-op | 7 | 5
  Post-op day 1: number analyzed (Participants) | 6 | 3
  Post-op day 1 | 6 | 3
  Post-op day 2: number analyzed (Participants) | 0 | 1
  Post-op day 2 | 0 | 1
  2 weeks post-op: number analyzed (Participants) | 5 | 3
  2 weeks post-op | 5 | 3
  3 weeks post-op: number analyzed (Participants) | 1 | 1
  3 weeks post-op | 1 | 1
  3 months post-op | 7 | 5
  6 months post-op: number analyzed (Participants) | 6 | 4
  6 months post-op | 6 | 4
  9 months post-op: number analyzed (Participants) | 1 | 0
  9 months post-op | 1 | 0
  1 year post-op: number analyzed (Participants) | 5 | 4
  1 year post-op | 5 | 4
  2 years post-op: number analyzed (Participants) | 0 | 1
  2 years post-op | 0 | 1

4. Secondary Outcome: Voice Quality After Total Thyroidectomy (TT) With and Without Prophylactic Central Neck Lymph Node Dissection (pCND) at 6 Months
Description: Participants that have improvement in voice quality after TT with and without pCND assessed by the Voice Handicap Index-10 questionnaire. The Voice Handicap Index-10 (VHI-10) is a self-administered questionnaire that assesses participant's subjective voice quality. The average voice scores/indices at 6 months post-operation was measured for all participants per group. Minimum score is 0 and maximum score is 40.The higher the score the worse voice quality.
Time Frame: baseline - pre-op and 6 months post-op
Population: One participant in Arm 2, and Arm 1 was inevaluable.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
score on a scale
  Baseline- Pre-op | 3 [0 to 13] | 0 [0 to 20]
  6 months Post-op | 3 [0 to 27] | 6 [0 to 25]

5. Secondary Outcome: Number of Participants With Hypoparathyroidism
Description: Number of participants with hypoparathyroidism 6 months post total thyroidectomy with and without prophylactic central neck lymph node dissection. Hypoparathyroidism occurs when one or more of your parathyroid glands are underactive and can lead to low parathyroid hormone and hypocalcemia.
Time Frame: 6 months
Population: One participant in Arm 2, and Arm 1 was inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
Participants | 2 | 5

6. Secondary Outcome: Number of Participants That Have Cervical Wound Complications
Description: number of participants that have cervical wound complications such as a hematoma, seroma, and/or surgical site infection.
Time Frame: 3 months
Population: One participant in Arm 2, and Arm 1 was inevaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
Participants
  Hematoma | 0 | 0
  Seroma | 0 | 0
  Surgical site infection | 0 | 0

7. Secondary Outcome: B-Raf Proto-oncogene Serine/Threonine Kinase (BRAF) Valine 600 Glutamic Acid (V600E) Mutation Status on Lymph Node Metastasis
Description: Correlation between BRAF V600E of tumor
Time Frame: At progression
Population: This outcome measure was not done because data were not collected.
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Proportion of Participants That Have Less Neck Pain.
Description: Proportion of participants that have less neck pain assessed by the Neck Pain Scale (0 = no pain, and 10 = unimaginable, unspeakable pain).
Time Frame: 6 months
Population: This outcome measure was not done because data were not collected.
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Improvement in Swallowing Impairment After Total Thyroidectomy (TT) With and Without Prophylactic Central Neck Lymph Node Dissection (pCND) at 6 Months
Description: Participants that have improvement in swallowing impairment after Total Thyroidectomy (TT) with and without Prophylactic Central Neck Lymph Node Dissection (pCND) assessed by the Swallowing Impairment Score (SIS-6) questionnaire. The average swallowing scores/indices at 6 months post-operation was measured for all participants per group. Minimum score is 0 and maximum score is 24. The higher the score indicates worse swallowing symptoms.
Time Frame: baseline - pre-op and 6 months post-op
Population: One participant in Arm 2, and Arm 1 was inevaluable.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
score on a scale
  Baseline - Pre-op | 0 [0 to 15] | 3 [0 to 6]
  6 months Post-op | 4 [0 to 19] | 5 [0 to 18]

10. Secondary Outcome: Number of Participants Who Developed Disease Progression or Recurrence After Surgery
Description: Disease progression is defined as a clinically detectable evidence of disease recurrence after surgery. Disease recurrence is the progression since participants were deemed to have no evidence of disease after surgery. Post-op ultrasounds were assessed for findings that are indicative/suspicious of disease recurrence. No specific response criteria (i.e. RECIST) was used. Ultrasound of neck soft tissue findings indicate progression/recurrence.
Time Frame: Completed at pre-operation (op), 3 months, 6 months, 1 year, 2 years and 3 years post-op.
Population: One participant in Arm 2, and two participants in Arm 1 was inevaluable. And not all participants in Arm 2 and Arm 1 had an ultrasound of the neck at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 7 | 5
Participants
  Pre-op | 0 | 0
  3 months | 0 | 0
  6 months: number analyzed (Participants) | 5 | 5
  6 months | 0 | 0
  1 year: number analyzed (Participants) | 5 | 5
  1 year | 0 | 0
  2 years: number analyzed (Participants) | 4 | 2
  2 years | 0 | 0
  3 years: number analyzed (Participants) | 1 | 1
  3 years | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 46 months and 23 days for the first group and 48 months and 3 days for the second group.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
Number analyzed (Participants) | 8 | 6
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 46 months and 23 days for the first group and 48 months and 3 days for the second group.
Arm/Group | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) | Arm 1/Total Thyroidectomy (TT) Alone
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 1/8 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2/Total Thyroidectomy (TT) Plus Prophylactic Central Neck Dissection (pCND) (N=8) | Arm 1/Total Thyroidectomy (TT) Alone (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT02408887/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/87/NCT02408887/ICF_001.pdf